CLINICAL TRIAL: NCT03334669
Title: Empowerment as a Mechanism for Change in Childhood Obesity Prevention
Brief Title: Family-centered Obesity Prevention: Communities for Healthy Living (CHL)
Acronym: CHL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The primary trial was halted due to covid-19 in the last 6 months of the trial; as a result, the intervention was not fully implemented and the final outcomes were not measured. Outcomes will be assessed with the data available (BL, Y1, Y2).
Sponsor: Boston College (Other)
Collaborators: Action for Boston Community Development (Other); Community Action Agency of Somerville (Unknown); Harvard School of Public Health (HSPH) (Other); University at Albany (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kirsten, Donahue and DiFelice Professor of Social Work, Boston College
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 15-3559
Record Dates: First submitted 2017-10-10; First posted 2017-11-07 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Pediatric Obesity; Obesity
Keywords: Childhood obesity; Preschool; Head Start; Family Interventions; Community Based Participatory Research (CBPR); Empowerment Theory; Family Ecological Theory; Step Wedge Design; Low Income
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Intervention Model Description: The stepped wedge design is a pragmatic design that is well suited for interventions that use a service delivery protocol and do not rely on individual recruitment of participants. The intervention is integrated into Head Start service delivery and data compiled for all enrolled children are used to evaluate the intervention. NOTE: Due to COVID-19 shutdown the final group of Head Start programs did receive the full intervention. The investigators elected to assess intervention impact with one year less data than expected. Due to low power, sensitivity analyses will examine the roles of dose, fidelity, baseline child overweight/obesity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Sites randomized to the intervention group will receive the following:
  1. Parents Connect for Healthy Living (PConnect)
  2. Enhanced Nutrition Support
  3. Media Resources
  Interventions: Behavioral: Parents Connect for Healthy Living (PConnect); Behavioral: Enhanced Nutrition Support; Behavioral: Media Resources
- Control (No Intervention): Control sites will not receive any intervention components (i.e., standard practice).

INTERVENTIONS:
Behavioral: Parents Connect for Healthy Living (PConnect) — Parents Connect for Healthy Living (PConnect) parent curriculum: This 10-week program (20 hours total) engages Head Start parents in a wide range of topics related to health and empowerment and is designed to foster a safe, open forum through which parents can connect with other parents and mobilize resources to support their family's health; NOTE: The PConnect program was not implemented in 2019-2020 due to the coronavirus pandemic. In 2020-2021, PConnect was implemented virtually; these are pilot data and not part of the main trial.
  Arms: Intervention
Behavioral: Enhanced Nutrition Support — Enhanced Nutrition Support: Existing nutrition resources within Head Start (e.g., Biannual child health letters) are expanded and improved to ensure parents are aware of their child's weight status and are linked with age-appropriate weight management services if their child has overweight or obesity. NOTE: Enhanced nutrition support was not implemented in spring 2020 due to the pandemic. In 2020-2021, it was moved to a virtual format in what will be a pilot virtual trial.
  Arms: Intervention
Behavioral: Media Resources — Media Resources: Print and online resources that employ consistent messaging to reach parents and ensure that behavior change messages are accessible to families. NOTE: Due to the pandemic, media resources were not shared in spring 2020. They were implemented in virtual format in 2020-2021 in a pilot virtual trial.
  Arms: Intervention

SUMMARY:
The Communities for Healthy Living (CHL) program is a family-focused intervention to promote healthy lifestyle behaviors including diet and physical activity among children (age 3-to 5-years) and their families, enrolled in Head Start.

DETAILED DESCRIPTION:
This evaluation will test the effectiveness of a family-focused intervention, Communities for Healthy Living (CHL), implemented through Head Start. Over 20% of preschool-aged children in the US experience overweight or obese. Because obesity prevention depends heavily on the adoption of healthy lifestyle behaviors early in life, preventive efforts offer a higher promise for success if they are family-centered. Effective family-centered interventions for obesity prevention in preschool-aged children, however, remain elusive. While a number of interventions have shown positive effects on child Body Mass Index (BMI), results are inconsistent and short term effects are not maintained. What is more, because families at greatest risk of childhood obesity - including low-income, single-parent, and ethnic minority families - are the most difficult to recruit and retain, results are often limited in their applicability to high risk populations.

In response, the researchers have partnered with Head Start to develop and test a new approach to family-centered childhood obesity prevention that addresses family engagement upfront. The CHL program will be refined and rigorously tested for efficacy in collaboration with Head Start programs in the greater Boston area, which collectively serve over 2000 low-income children each year. Building on a previous pilot study, the investigators will broaden the parent-centered Community Based Participatory Research approach and include Head Start staff in the decision making and implementation process, refine intervention components, and expand technical assistance protocols to support Head Start ownership of CHL while ensuring implementation fidelity. In addition, consistent with the overarching theoretical framework (Family Ecological Model), neighborhood-level socioeconomic, food and physical activity environments around family homes and examine their impact on intervention outcomes will be measured to inform future scale up efforts.

ELIGIBILITY:
Primary Outcome Measures

Inclusion:

* Enrolled in a participating Head Start program
* Age 33 months to 5 years (i.e., meets Head Start age eligibility criteria)

Exclusion:

* Those not meeting inclusion criteria

Secondary Outcome Measures

Inclusion:

* Enrolled in a participating Head Start program
* Age 33 months to 5 years

Exclusion:

* Children not enrolled at a participating Head Start program
* Children less than 29 months or older than 59 months by Sept 1

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4999 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Child BMI-z score | Collected at the beginning and end of each academic year (i.e., fall, spring) for 3 years (BL, Y1, Y2) rather than 4 years as planned
  Change in child BMI-z score
Modified change in BMI z-score | Collected at the beginning and end of each academic year (i.e., fall, spring) for 3 years (BL, Y1, Y2)
  BMI of a child is expressed relative to the median BMI in units of ½ of the distance between 0 and +2 z- scores. https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5703793/

SECONDARY OUTCOMES:
Change in child fruit and vegetable intake | Collected at the beginning and end of each academic year (i.e., fall, spring) for 3 years (BL, Y1, Y2) rather than 4 years as planned
  Change in child fruit and vegetable intake assessed by parent report of child weekly frequency of intake
Change in child sugar-sweetened beverage intake | Collected at the beginning and end of each academic year (i.e., fall, spring) for 3 years (BL, Y1, Y2) rather than 4 years as planned
  Change in child sugar-sweetened beverage consumption assessed by parent report of child weekly frequency of intake
Change in child physical activity | Collected at the beginning and end of each academic year (i.e., fall, spring) for 3 years (BL, Y1, Y2) rather than 4 years as planned
  Change in child physical activity assessed by parent report of average minutes per day child spent in structured free play and organized physical activities
Change in child sleep duration | Collected at the beginning and end of each academic year (i.e., fall, spring) for 3 years (BL, Y1, Y2) rather than 4 years as planned
  Change in child daily sleep duration assessed by parent report (calculated from average bedtime and wake time)
Change in child screen-time | Collected at the beginning and end of each academic year (i.e., fall, spring) for 3 years (BL, Y1, Y2) rather than 4 years as planned
  Change in child daily hours of screen-time exposure (TV, computer, tablet) assessed by parent completion of the School Physical Activity and Nutrition Survey (SPAN)
Summer weight gain | Summer weight gain was assessed over 3 summer periods using BMI data collected at the beginning and end of each academic year
  Change in child BMIz (and modified BMIz) over the summer period

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Davison, PhD, Principal Investigator — Boston College
Locations (1):
- Boston College, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leipner N, Liesenfeld H. [Synchronous bilateral testicular tumor: embryonal carcinoma and Leydig cell tumor]. Aktuelle Radiol. 1995 May;5(3):179-80. German. PMID 7605818
- [Background] Thomson AB, Babiuk L, Kirdeikis P, Zuk L, Marriage B, Bowes K. A dose-ranging study of ranitidine and its effect on intragastric and intra-oesophageal acidity in subjects with gastro-oesophageal reflux disease. Aliment Pharmacol Ther. 1994 Aug;8(4):443-51. doi: 10.1111/j.1365-2036.1994.tb00312.x. PMID 7986969
- [Background] Guler N, Yalcin I, Salman N, Ones U. Invasive pulmonary aspergillosis in chronic granulomatous disease: response to systemic prednisolone treatment and locally applied amphotericin B. Turk J Pediatr. 1994 Oct-Dec;36(4):341-5. PMID 7825243
- [Background] Shaw NA. The effects of electroconvulsive shock on the thalamic auditory potential. Biol Psychiatry. 1996 Oct 15;40(8):807-10. doi: 10.1016/0006-3223(96)00252-1. No abstract available. PMID 8894077
- [Background] Ries JC, Schreiner D, Steininger H, Girod SC. p53 mutation and detection of p53 protein expression in oral leukoplakia and oral squamous cell carcinoma. Anticancer Res. 1998 May-Jun;18(3B):2031-6. PMID 9677462
- [Background] Kesselring A. [Opening address. Family caregivers: what challenges for the future?]. Krankenpfl Soins Infirm. 2001 Jul;94(7):18-21. No abstract available. German. PMID 11944454
- [Background] Delahaye L, Mothe-Satney I, Myers MG, White MF, Van Obberghen E. Interaction of insulin receptor substrate-1 (IRS-1) with phosphatidylinositol 3-kinase: effect of substitution of serine for alanine in potential IRS-1 serine phosphorylation sites. Endocrinology. 1998 Dec;139(12):4911-9. doi: 10.1210/endo.139.12.6379. PMID 9832428
- [Background] Beckerman JP, Aftosmes-Tobio A, Kitos N, Jurkowski JM, Lansburg K, Kazik C, Gavarkovs A, Vigilante A, Kalyoncu B, Figueroa R, Klabunde R, Barouch R, Haneuse S, Taveras E, Davison KK; CHL study team. Electronic address: chlheadstart@gmail.com. Communities for healthy living (CHL) - A family-centered childhood obesity prevention program integrated into Head Start services: Study protocol for a pragmatic cluster randomized trial. Contemp Clin Trials. 2019 Mar;78:34-45. doi: 10.1016/j.cct.2019.01.002. Epub 2019 Jan 7. PMID 30630109
- [Background] Beckerman-Hsu JP, Aftosmes-Tobio A, Gavarkovs A, Kitos N, Figueroa R, Kalyoncu ZB, Lansburg K, Yu X, Kazik C, Vigilante A, Leonard J, Torrico M, Jurkowski JM, Davison KK. Communities for Healthy Living (CHL) A Community-based Intervention to Prevent Obesity in Low-Income Preschool Children: Process Evaluation Protocol. Trials. 2020 Jul 23;21(1):674. doi: 10.1186/s13063-020-04571-0. PMID 32703293
- [Derived] Gago C, Aftosmes-Tobio A, Beckerman-Hsu JP, Oddleifson C, Garcia EA, Lansburg K, Figueroa R, Yu X, Kitos N, Torrico M, Leonard J, Jurkowski JK, Mattei J, Kenney EL, Haneuse S, Davison KK. Evaluation of a cluster-randomized controlled trial: Communities for Healthy Living, family-centered obesity prevention program for Head Start parents and children. Int J Behav Nutr Phys Act. 2023 Jan 11;20(1):4. doi: 10.1186/s12966-022-01400-2. PMID 36631869
- [Derived] Grafft N, Aftosmes-Tobio A, Gago C, Lansburg K, Beckerman-Hsu J, Trefry B, Kumanyika S, Davison K. Adaptation and implementation outcomes of a parenting program for low-income, ethnically diverse families delivered virtually versus in-person. Transl Behav Med. 2022 Nov 21;12(11):1065-1075. doi: 10.1093/tbm/ibac077. PMID 36318233
- [Derived] Beckerman-Hsu JP, Gago C, Aftosmes-Tobio A, Jurkowski JM, Lansburg K, Leonard J, Torrico M, Haneuse S, Subramanian SV, Kenney EL, Davison KK. Acceptability and appropriateness of a novel parent-staff co-leadership model for childhood obesity prevention in Head Start: a qualitative interview study. BMC Public Health. 2021 Jan 22;21(1):201. doi: 10.1186/s12889-021-10159-3. PMID 33482774